CLINICAL TRIAL: NCT05048745
Title: Recurrent Appendicitis Following Successful Drainage of Appendicular Abscess in Adult Without Interval Appendectomy During COVID-19. Prospective Cohort Study
Brief Title: Recurrent Appendicitis Following Successful Drainage of Appendicular Abscess in Adult
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer Alsaied Alnaimy, assistant professour of general and laparoscopic surgery, Zagazig University
Other Study IDs: recurrent appendicitis
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Appendicitis
Keywords: appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: interval appendectomy — interval appendectomy

SUMMARY:
COVID-19 infection is a global pandemic that locked down hospitals and made patients fear to consult for medical health problems especially acute abdominal pain. Subsequently, complicated appendicitis namely appendicular abscess in increasing. The best treatment of an appendicular abscess is percutaneous drainage while no studies are dealing with recurrent appendicitis in cases without interval appendectomy during the COVID-19 pandemic. This study aimed to evaluate recurrent appendicitis after successful drainage of appendicular abscess without interval appendectomy during COVID.

A prospective cohort study conducted in the surgical emergency units of University Hospitals between 15th March 2020 to 15th August 2020 on 316 patients admitted during the study period with the clinical diagnosis of a successful drained appendicular abscess. (Open or radiological).

DETAILED DESCRIPTION:
The novel coronavirus SARS-CoV-2 (causing COVID-19) was first discovered in Wuhan in China at the end of 2019 then at the beginning of 2020, World Health Organization (WHO) announced COVID-19 as a global pandemic [1]. Because the virus is highly infectious, hospitals all over the world became overloaded by COVID-19 infected patients, and a state of emergency is announced and the population was advised to stay at home. Moreover, people were afraid to become infected by the virus and hence there is marked reductions in consultation of medical advice even the acute abdominal cases. [2-3] Acute appendicitis is the commonest cause of acute abdomen in all ages with an incidence risk of 7%-8% worldwide [4]. Complicated appendicitis represents nearly4%-25% of cases [5]. Appendicular abscess formation occurs in 2-7% of patients with perforated appendicitis [6]. Delay in medical consultation is a leading cause for developing complicated appendicitis [5]. In patients with an appendicular abscess, a non-operative treatment, with ultrasonography of computerized tomography (CT) guided drainage and antibiotic treatment is starting initially and then interval appendectomy is performed later. This approach lowers the peri- and postoperative complications [7-10].

Surgeons preferring interval appendectomy have a concept that the incidence of recurrence of appendicitis is high and by performing interval appendectomy the underlying pathology like Crohn's disease or malignancy cannot be missed and dealt with in time [11]. Others have opposed this concept as the reported incidence of recurrent appendicitis is ranges from 3.4% to 25.5%, with the greatest risk during the first 3 months after the initial episode [12-13]. The aim was evaluating recurrence appendicitis (the true incidence, rate, severity , and risk factors) in patients treated without interval appendectomy in cases following successful drainage of appendicular abscess during the pandemic of COVID-19. Previous studies handled recurrent appendicitis but non-complicated patients, however, Up to our knowledge, no study handled the actual recurrence rates severity, and risk factors in non-operative treatment of complicated appendicitis with abscess during the COVID-19 pandemic.

2. Material and Methods: 3.1 Study design and setting: Prospective cohort study conducted in the surgical emergency units of University Hospitals between 15th March 2020 to 15th August 2020 on 316 patients admitted during the study period with the clinical diagnosis of a successful drained appendicular abscess. (Open or radiological). This study is compliant with the STROCSS criteria [14].

3.2 Patient selection: Inclusion criteria included age >16 years, both sex and successful drained appendicular abscess while exclusion criteria included patients 16≤ years, generalized peritonitis, pregnancy, cases suspected of cancer caecum, inflammatory bowel disease, failure or difficult initial drainage e.g. pelvic abscess, appendectomy performed at the time of drainage, non-cooperative patients for regular follow up and abscess less than 3 cm if showed improvement of clinical and radiological signs within 3 days of antibiotic therapy alone.

3.3 Types of outcome measures: The outcomes were incidence, severity, and risk factors of recurrence appendicitis in patients without interval appendectomy (clinical or radiological at any time point during follow up period).

3.4 Outcomes measurement: The diagnosis of the appendicular abscess was based on presentation with right lower quadrant abdominal pain, fever, palpable or suspicion of a mass with tenderness. The presence of abscess was confirmed in all patients by ultrasound (US) or computed tomography (CT) scan. Morbidity and mortality were evaluated by Dindo and Clavien classification [15]. Successful drainage was detected by the absence of symptoms and normalization of laboratory and radiological investigation (WBCs and sonar). Recurrent appendicitis was diagnosed if recurrent abdominal pain was associated with tenderness/ rebound tenderness with or without fever. The severity of recurrent appendicitis is measured by a score [16].

3.5 Procedure: appendectomy was performed either by open approach (77.1% of cases) or laparoscopic approach in the remaining cases. Steps of operations were according to ordinary steps described in the previous study [17]. All appendixes were examined histologically.

3.6 discharge and follow up parameters Following successful drainage of appendicular abscess, Patients were discharged from the hospital when normalization of white blood cell count (below 12,000 cells/mm3), absent fever, no abdominal pain nor tenderness, and ability to tolerate oral intake. Patients were typically discharged on oral antibiotics for a week in the form of third-generation cephalosporin and metronidazole. Those discharged from the hospital were followed up in an outpatient department monthly for the first three months, and once every three months for the following nine months. During the outpatient interviews, all patients were clinically examined. Colonoscopy and CT were performed routinely on patients above the age of 40years. Patients with recurrent symptoms of appendicitis were offered appendectomy. The patients not attending the outpatient visit were also contacted by telephone or e-mail to obtain information on their status.

Our study evaluated recurrent appendicitis(incidence, rate, severity and risk factors) after successful drainage of appendicular abscess without interval appendectomy during one year follow up in the era of COVID-19 when there is a global tendency for postponing non-emergent surgeries. One of these cases was interval appendectomy following drainage of an appendicular abscess.

Although previous studies handled recurrent appendicitis following successful drainage of an appendicular abscess but these studies were performed before the era of COVID-19, while, other studies faced recurrent appendicitis in the era of COVID-19 with non-operative treatment but in non-complicated appendicitis. Yet, no studies faced recurrent appendicitis following complicated appendicitis drainage in the era of COVID-19. Based on our results, we found that recurrent appendicitis occurred in 30.4% of cases underwent successful drainage of appendicular abscess during 1 year follow up during COVID-19, and 43.7% of them, recurrence occurred within the first 3 months after drainage and 56.3% of them showed recurrence after 3 month up to 1 year. Incidence of recurrent appendicitis is high in our results and this is attributed to the fact that COVID-19 induces vasculitis and thrombotic occlusion of the appendicular artery. Furthermore, COVID-19 causes hyperplasia of lymphoid tissue in the wall of the appendix causing an obstruction. Kaplan-Meier curve (Fig 2) confirmed that the rate of recurrent appendicitis is 13.3% in the first 3 months; then, later, the rate of recurrent appendicitis increased reaching up to 30% at one year follow up. So, we recommend performing interval appendectomy that will prevent recurrent appendicitis in 56.3% of cases of recurrent appendicitis and prevent the high rate of recurrent appendicitis after 3rd month.

Incidence of recurrent appendicitis varies between studies that may be as low as 8.9% [7] and 13% in a recent study published just before COVID-emergency [18] up to 27% in a third study[19]. Our study showed a higher recurrence rate (30.4%) that was most probably due to infection with covid-19. A study by Lai et al., [11] stated that the rate of appendicitis recurrence after conservative treatment was 25.5%; most recurred within 6 months after discharge (83.3%). The benefit of preventing recurrence is less than 16% if interval appendectomy is performed 6 weeks after discharge and less than 10% if it is done 12 weeks later. Another prospective study revealed that in¬terval appendectomy done at 6 and 12 weeks had prevent¬ed 10.6% and 6.7% of recurrent appendicitis respectively [20] which means that in 89.4% and 93.3% the interval ap¬pendectomy done was unnecessary. Our study showed that interval appendectomy could prevent 56.3% of recurrent appendicitis after 3 months (which is higher than the previous study). Infection with COVID-19 is the probable cause of a high incidence of recurrent appendicitis after 3 months. Before conducting our study, we thought that recurrent appendicitis during COVID-19 would be greater in severity. This thought was logical due to vasculitis and lymphoid hyperplasia, but the opposite result we found. We found that although the incidence of recurrent appendicitis is high, however, most cases were low in severity (63.5% grade I).Other studies agreed with this results in that severity of appendicitis is less in covid-19 [21-22]. We failed to explain this finding.

In our centers, laparoscopic appendectomy is the method of choice in treating acute appendicitis. However, during the era of covid-19; this trend was changed in our hospitals for fear of aerosol-induced transmission of covid-19 infection. most cases of recurrent appendicitis(77.1%) operated by open appendectomy. this attitude was approved by many studies [23-27] While another study [28] did not approve this consent and confirmed that the risks of laparoscopy are less than its benefits. Subsequently, our result showed that intraoperative complications occurred in 7.3% of cases mostly bleeding cystic artery while postoperative complications occurred in 15.6% of cases.

During covid-19, it is of profound importantance to detect risk factors and predictors of recurrent appendicitis during follow-up period. These patients are at great risk and interval appendectomy is intended for those patients. These predictors are older age (ASA III), abscess size > 3cm, and diabetes mellitus. Older age patients are susceptible to covid-19 infection due to decreased immunity especially if associated with other co-morbidities as D.M and hypertension. Older age is associated with atherosclerosis of the appendicular artery and atherosclerosis developed earlier in diabetic patients. A study that faced risk factors for recurrent appendicitis [13] stated that by using Cox regression, sex had a slight influence on recurrent appendicitis (hazard ratio males vs. females=0.52, 95% CI, 0.27- 0.99, P=.05). Age, Charlson comorbidity index, type of appendicitis, or percutaneous abscess drainage did not influence recurrence.

ELIGIBILITY:
Inclusion Criteria:

* both sex
* successful drained appendicular abscess

Exclusion Criteria:

* generalized peritonitis
* pregnancy
* cases suspected of cancer caecum, inflammatory bowel disease, failure or difficult initial drainage e.g. pelvic abscess, appendectomy performed at the time of drainage, non-cooperative patients for regular follow up and abscess less than 3 cm if showed improvement of clinical and radiological signs within 3 days of antibiotic therapy alone.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Prospective cohort study conducted in the surgical emergency units of our University Hospitals between 15th March 2020 to 15th August 2020 on 316 patients admitted during the study period with the clinical diagnosis of a successful drained appendicular abscess. (Open or radiological). This study is compliant with the STROCSS criteria
Sampling Method: Non-Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
recurrence | 1 year
  incidence of recurrence

CONTACTS AND LOCATIONS:
Overall Officials: tamer alnaimy, Phd, Principal Investigator — faculty of medicine zagazig university
Locations (1):
- Tamer Alsaied Alnaimy, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No